CLINICAL TRIAL: NCT02213198
Title: Improving Transitional Care Experiences in Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IH-1304-6506
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2016-11

CONDITIONS: Standard Treatment Versus Engagement Focused Treatment
Keywords: Serious mental illness transitions shared decision making
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Engagement Focused Care (Experimental): Engagement Focused Care which includes all components of standard treatment plus both group Access intake process with its flexibility of scheduling and the SDM intervention
  Interventions: Behavioral: Engagement focused care
- Standard Care (Active Comparator): Standard Care includes individual intake appointments which are traditional in outpatient service and all services of the clinic including counseling, access to a prescriber, care coordination, and access to home visits.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Engagement focused care — Engagement focused care includes a group intake appointment called Access group with flexible scheduling allowing ease of rescheduling and access as soon as the same day, as well as Shared Decision Making coaching. For Shared Decision Making, a coach meets with the person prior to or following appointments with the prescriber to assist the person regarding what to ask, what to tell, to review options, and to foster choice.
  Arms: Engagement Focused Care
Behavioral: Standard Care — Standard treatment provided by a university based transitional care clinic, with individual intakes and follow-ups for medication/therapy scheduled as soon as possible from intake but at least 1 week away-no prioritization of cases
  Arms: Standard Care

SUMMARY:
The cost of serious mental illness (SMI) in the U.S. is $317 billion annually. This translates to more than $1000 for every man, women, and child in the U.S. Hospitalization and Emergency Room (ER) visits have the highest costs. Outpatient services are overburdened. There is a push to get people out of hospitals quickly, while they are still quite ill. These factors cause patients to be lost in the transition from inpatient to outpatient care. Many individuals are repeatedly rehospitalized or continue to clog emergency rooms in an attempt to receive care. The importance of transitional care between inpatient/ER facilities and outpatient services to prevent this revolving door phenomenon has been continually stressed. There is little research on the best way to accomplish smooth transition to outpatient care. We developed a 90-day transitional care clinic (TCC) to address this need. We propose a randomized treatment outcome study comparing two transitional service packages within our TCC: a Standard Care package versus an Engagement-Focused package that features a novel intake procedure and a Shared Decision-Making intervention: Access Group is an intake procedure designed to address many of the problems of traditional approaches to post-acute treatment engagement, including failure of patients to reach intake appointments. Shared Decision-Making (SDM) is a structured approach to provider-patient communication that has been shown to increase patient involvement in care and improve outcomes. Despite SMI patients' desire to be more involved in their treatment decisions and promising early evidence of SDM's effectiveness in SMI, SDM has not been systematically evaluated in transitional psychiatric care. In the proposed study, patients referred to TCC will be randomized to either Engagement-focused Care or Standard Care. The relative benefit of these two approaches will be evaluated in 300 individuals who will be randomized to these two treatments in a 2:1 ratio. We hypothesize that attendance at appointments, reported satisfaction, shared decision making and quality of life will be higher for engagement focused care. The new treatment package is designed to get individuals into treatment quickly and to teach them how to be good consumers of mental health treatments going forward.

DETAILED DESCRIPTION:
Aim 1: To compare EFC to SC with respect to linkage to TCC services. Hypothesis A: Patients referred to EFC will exhibit a significantly greater rate of attendance at their TCC intake appointment than SC patients.

Aim 2: To compare EFC to SC with respect to patient participation in outpatient treatment.

Hypothesis B: Patients referred to EFC will report significantly greater shared decision-making in their TCC prescriber appointments than SC patients.

Hypothesis C: Patients referred to EFC will exhibit significantly greater attendance at post-intake scheduled TCC appointments than SC patients.

Hypothesis D: Patients referred to EFC will exhibit a significantly greater rate of attendance at initial post-TCC scheduled mental health appointments than SC patients.

Aim 3: To compare Engagement-focused Care (EFC) to Standard Care (SC) with respect to patients' long term quality of life.

Hypothesis E: Patients who receive EFC will exhibit significantly greater quality of life than SC patients six months after TCC termination.

ELIGIBILITY:
Inclusion Criteria:

* Serious mental illness including (schizophrenia, schizoaffective disorder, mood disorders, anxiety disorders), referral from inpatient psychiatric unit or emergency service at the time of discharge to the Transitional Care Clinic, ability to sign informed consent

Exclusion Criteria:

* Unable to complete assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I Velligan, PhD, Principal Investigator — University of Texas
Locations (1):
- UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data provided by PI as requested velligand@uthscsa.edu

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Engagement Focused Care | Standard Care
Started | 306 | 159
Completed | 218 | 108
Not Completed | 88 | 51
Not completed — No show for intake | 7 | 9
Not completed — Withdrawal by Subject | 34 | 11
Not completed — transferred out of clinic | 7 | 9
Not completed — Lost to Follow-up | 40 | 21
Not completed — incarcerated,violent | 0 | 1
Period: Follow up 1 3 Mos Post BL End of TCC tx
Arm/Group | Engagement Focused Care | Standard Care
Started | 218 | 108
Completed | 125 | 67
Not Completed | 93 | 41
Not completed — Withdrawal by Subject | 4 | 4
Not completed — rehab/incarceration/violence | 3 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 68 | 25
Not completed — unable to contact at 3 but got 6 post DC | 17 | 10
Period: Follow up 2 6 Months Post TCC Treatment
Arm/Group | Engagement Focused Care | Standard Care
Started | 125 | 67
Completed | 102 | 60
Not Completed | 23 | 7
Not completed — Lost to Follow-up | 23 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engagement Focused Care | Standard Care | Total
Number analyzed (Participants) | 219 | 107 | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 219 | 107 | 326
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (11.4) | 39.9 (13.1) | 38 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 56 | 179
  Male | 96 | 51 | 147
Region of Enrollment [Number; unit: participants]
  United States | 219 | 107 | 326

OUTCOME MEASURES:

1. Primary Outcome: Subjective Quality of Life
Description: The Quality of Life Interview (QOLI; 91) is a 45-minute structured interview that assesses quality of life in the domains of family, social relations, leisure activities, finances, legal/safety issues, work/school, and health. It is one of the most psychometrically sound QoL instruments for use in mental illness. The subjective scale assesses quality of life from the perspective of the patient. Subjective QOL = Mean of items 1,3,8,9,11,13,16,18,20,21 . Scores range from 1-7. Higher scores indicate better quality of life
Time Frame: baseline, 3 months and 6 months
Population: All patients with baseline and at least one follow up on QOL
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engagement Focused Care | Standard Care
Number analyzed (Participants) | 219 | 107
units on a scale
  Baseline | 3.9 (1.1) | 3.8 (1.1)
  TCC Discharge at 3 months | 4.3 (1.1) | 4.0 (1.0)
  Follow up 6 mos post TCC | 4.5 (1.1) | 4.2 (1.0)

2. Primary Outcome: Engagement in Treatment
Description: Whether patient kept appointment post TCC
Time Frame: 6 months
Population: All patients for whom survey (call data) were available post TCC discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement Focused Care | Standard Care
Number analyzed (Participants) | 124 | 69
Participants | 78 | 40

ADVERSE EVENTS:
Time Frame: 9-12 months
Arm/Group | Engagement Focused Care | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/306 | 0/159
Other Adverse Events (participants affected / at risk) | 0/306 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No